CLINICAL TRIAL: NCT02135679
Title: The Detection Of Circulating Tumor Cells (CTC) In Patients With Non-small Cell Lung Cancer (NSCLC) Undergoing Definitive Radiotherapy Or Chemoradiotherapy
Brief Title: The Detection Of Circulating Tumor Cells (CTC) In Patients With NSCLC Undergoing Definitive Radiotherapy Or Chemoradiotherapy
Status: Completed | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 12512
Record Dates: First submitted 2014-05-02; First posted 2014-05-12 (Estimated); Results first posted 2024-10-08 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (7):
- Cohort 1: Patients with early stage NSCLC undergoing stereotactic radiotherapy
  Interventions: Radiation: Radiotherapy
- Cohort 2: Patients with locally advanced NSCLC undergoing standard chemoradiotherapy
  Interventions: Radiation: Radiotherapy
- Cohort 3: Patients with stage I-III NSCLC undergoing standard, fractionated radiotherapy alone
  Interventions: Radiation: Radiotherapy
- Cohort 4: Patients with locally advanced NSCLC undergoing standard chemoradiotherapy with the novel signal transduction inhibitor, nelfianvir.
  Interventions: Radiation: Radiotherapy
- Cohort 5: Patients with resectable stage IIIa NSCLC undergoing pre-operative chemoradiotherapy
  Interventions: Radiation: Radiotherapy
- Cohort 6: Patients with suspected (no tissue diagnosis) early stage NSCLC undergoing stereotactic radiotherapy
  Interventions: Radiation: Radiotherapy
- Cohort 7: Patients with locally advanced NSCLC undergoing stereotactic radiotherapy followed by concurrent mediastinal chemoradiotherapy
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Radiation: Radiotherapy

SUMMARY:
CTC levels collected pre-surgery will be correlated with pathological samples.

DETAILED DESCRIPTION:
Patients with NSCLC who undergo radiation as part of a definitive course of treatment will be enrolled. Blood collections will be obtained before, during, and after radiotherapy. We will collect demographic and treatment data and explore & describe the pattern of CTC detection in all patients

ELIGIBILITY:
Inclusion Criteria:

* Patients with biopsy-proven NSCLC who are undergoing definitive radiotherapy as a part of their treatment regimen.
* Age 18 or older
* Signed informed consent
* Patients who are incapable of providing informed consent are excluded from participating in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: NSCLC patients
Sampling Method: Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2012-09; Primary Completion 2019-12 (Actual); Study Completion 2021-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Feigenberg, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Evanson D, Griffin M, O'Reilly SE, Johnson T, Werner T, Kothekar E, Jahangiri P, Simone CB 2nd, Swisher-McClure S, Feigenberg SJ, Revheim ME, Zou J, Alavi A. Comparative assessment of radiation therapy-induced vasculitis using [18F]FDG-PET/CT in patients with non-small cell lung cancer treated with proton versus photon radiotherapy. Eur J Nucl Med Mol Imaging. 2024 Apr;51(5):1444-1450. doi: 10.1007/s00259-023-06535-3. Epub 2023 Dec 14. PMID 38095673

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Patients with early stage NSCLC undergoing stereotactic radiotherapy
  Radiotherapy
- Cohort 2: Patients with locally advanced NSCLC undergoing standard chemoradiotherapy
  Radiotherapy
- Cohort 3: Patients with stage I-III NSCLC undergoing fractionated radiotherapy alone
  Radiotherapy
- Cohort 4: Patients with locally advanced NSCLC undergoing standard chemoradiotherapy with the signal transduction inhibitor, nelfianvir.
  Radiotherapy
- Cohort 5: Patients with resectable stage IIIa NSCLC undergoing pre-operative chemoradiotherapy
  Radiotherapy
- Cohort 6: Patients with suspected (no tissue diagnosis) early stage NSCLC undergoing stereotactic radiotherapy
  Radiotherapy
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7
Started | 52 | 69 | 2 | 0 | 18 | 63 | 0
Completed | 39 | 51 | 1 | 0 | 16 | 57 | 0
Not Completed | 13 | 18 | 1 | 0 | 2 | 6 | 0

BASELINE CHARACTERISTICS:
Population: There was no eligible participant for cohort 4 and cohort 7
Groups:
- Cohort 4: Patients with locally advanced NSCLC undergoing standard chemoradiotherapy with the signal transduction inhibitor, nelfianvir
  Radiotherapy
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7 | Total
Number analyzed (Participants) | 52 | 69 | 2 | 0 | 18 | 63 | 0 | 204
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 24 | 1 | 0 | 10 | 13 | 0 | 56
  >=65 years | 44 | 45 | 1 | 0 | 8 | 50 | 0 | 148
Age, Continuous [Median (Full Range); unit: years] | 75 [59 to 93] | 66 [31 to 84] | 68 [58 to 78] |  | 63.5 [29 to 80] | 70 [55 to 91] |  | 69 [29 to 93]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 35 | 2 | 0 | 6 | 33 | 0 | 107
  Male | 21 | 34 | 0 | 0 | 12 | 30 | 0 | 97
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Black or African American | 10 | 14 | 0 | 0 | 2 | 12 | 0 | 38
  White | 39 | 53 | 2 | 0 | 15 | 49 | 0 | 158
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 52 | 69 | 2 | 0 | 18 | 63 | 0 | 204
Biopsy-Proven Non-Small Cell Lung Cancer [Count of Participants; unit: Participants] | 52 | 69 | 2 | 0 | 18 | 0 | 0 | 141

OUTCOME MEASURES:

1. Primary Outcome: To Describe the Pattern of CTCs Before and After Definitive Radiotherapy for Each Treatment Stratum
Description: The pattern of CTCs before and after definitive radiotherapy for each treatment stratum. CTC counts per mL before and after definitive radiotherapy.
Time Frame: 24 months
Population: There were no enrolled patients in Cohorts 4 and 7. The Overall Number of Participants Analyzed in the Arms/Groups is not consistent with numbers provided in the Participant Flow module because not all patients underwent sequential (multiple) assays necessary for analysis. Only 114 out of 204 patients fulfilled the analysis criteria such as sequential PET/CT scans performed in the home institution.
Measure: Median (Full Range); unit: CTCs/mL
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7
Number analyzed (Participants) | 21 | 50 | 2 | 0 | 6 | 35 | 0
CTCs/mL
  CTC counts per mL before definitive radiotherapy. | 3.9 [0 to 209] | 9.1 [0.57 to 570.7] | 9.1 [0.57 to 570.7] |  | 9.1 [0.57 to 570.7] | 3.9 [0 to 209] |
  CTC counts per mL after definitive radiotherapy. | 0.4 [0 to 5.5] | 0.6 [0 to 1.8] | 0.6 [0 to 1.8] |  | 0.6 [0 to 1.8] | 0.4 [0 to 5.5] |

ADVERSE EVENTS:
Time Frame: Adverse events were not followed or reported for this protocol.
Description: Adverse events were not followed or reported for this protocol.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-02): https://cdn.clinicaltrials.gov/large-docs/79/NCT02135679/Prot_SAP_000.pdf